CLINICAL TRIAL: NCT02822612
Title: A Prospective Single-Site Non-Interventional Study to Evaluate Human Factors and Usability of Automated, Comprehensive Ocular Examination in Elderly and Visually Impaired Populations Using a Prototype Binocular Optical Coherence Tomography System
Brief Title: The EASE Study - Human Factor and Usability Testing of a Binocular OCT System
Acronym: EASE
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/LO/1756
Record Dates: First submitted 2016-06-23; First posted 2016-07-04 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Glaucoma; Retinal Disease; Strabismus; Healthy Volunteers
Keywords: optical coherence tomography; optical imaging; retinal imaging
MeSH Terms: conditions — Glaucoma; Retinal Diseases; Strabismus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Retinal Disease: Fifteen subjects with retinal disease. Each participant will attend for a single study visit, lasting approximately 1 hour in duration.
  Interventions: Device: Binocular OCT prototype
- Glaucoma: Fifteen subjects with glaucoma. Each participant will attend for a single study visit, lasting approximately 1 hour in duration.
  Interventions: Device: Binocular OCT prototype
- Strabismus: Fifteen subjects with strabismus. Each participant will attend for a single study visit, lasting approximately 1 hour in duration.
  Interventions: Device: Binocular OCT prototype
- Healthy volunteers: Fifteen healthy volunteers. Each participant will attend for a single study visit, lasting approximately 1 hour in duration.
  Interventions: Device: Binocular OCT prototype

INTERVENTIONS:
Device: Binocular OCT prototype — Testing will begin using a prototype binocular OCT system. Subjects will undergo the full suite of diagnostic assessments offered by the system at that time (i.e., visual acuity, ophthalmic history, pupillometry, ocular motility, perimetry, anterior segment and posterior segment OCT imaging).

SUMMARY:
Ophthalmology is among the most technology driven of all medical specialties, with advanced medical imaging devices - and specialised computer software - increasingly adopted for routine clinical use. While many such devices are capable of completing specific tasks, lack of "usability" prevents their widespread adoption (i.e., such devices are not easy to learn and remember, or are not efficient or subjectively pleasing to use). Moreover, devices that are difficult to use expose patients to clinical risk as a result of human error during usage.

With the introduction of a new medical technology, it is essential, therefore, to have a deep understanding of patients, what they need, what they value, their abilities, and also their limitations.

Human factor and usability testing, also known as "human factor engineering", deals with the formal study of people's interaction with their environment (in this case, the binocular optical coherence tomography (OCT) device). Structured, patient-centred, usability testing is essential to the design, clinical validation, regulatory approval, and widespread implementation, of all new medical devices. This is particularly the case for a putative binocular OCT system - a device intended for automated use in visually impaired, often elderly, populations. Although the binocular OCT is already at an advanced stage of hardware development, the EASE study will facilitate an iterative process of operating software and workflow modifications to optimize the device for use in these populations.

ELIGIBILITY:
Inclusion criteria for participants with chronic eye disease will include:

* Presence of retinal disease, glaucoma or strabismus
* Male or female, aged 18 years or older
* Ability to understand nature/purpose of the study and to provide informed consent
* Ability to undergo binocular OCT imaging
* Ability to follow instructions and complete the study
* Ability to speak English

Exclusion criteria for participants with chronic eye disease will include:

* Optical media opacity sufficient to preclude adequate ocular imaging with OCT
* Hearing impairment sufficient to interfere with hearing instructions
* Any condition which, in the investigator's opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule, or other study conduct.

Inclusion criteria for healthy subjects will include:

* No self-reported ocular history (although wearing corrective prescription glasses is permitted)
* Male or female, aged 18 years or older
* Ability to understand nature/purpose of the study and to provide informed consent
* Ability to undergo binocular OCT imaging
* Ability to follow instructions and complete the study
* Ability to speak English

Exclusion criteria for healthy subjects will include:

* Presence of ocular pathology
* Hearing impairment sufficient to interfere with hearing instructions
* Any condition which, in the investigator's opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule, or other study conduct.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with chronic eye disease (retinal disease, glaucoma, and strabismus) will be recruited from appropriate eye clinics at Moorfields Eye Hospital and from a patient advisory group established for this purpose.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS FT, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Retinal Disease: Fourteen participants had bilateral retinal disease only (including 8 with age-related macular degeneration [AMD], 4 with diabetic macular edema, 1 with central serous retinopathy, and 1 with retinal vein occlusion with cystoid macular edema).
- Glaucoma: Thirteen participants had glaucoma only (12 with primary open angle glaucoma [POAG], 1 with glaucoma secondary to hypertensive uveitis).
- Strabismus: Fourteen participants had strabismus only (7 with esotropia, 6 with exotropia, and 1 with hypertropia).
- Ocular Comorbidities: Four participants had ocular comorbidities: two with bilateral POAG and AMD; one had unilateral POAG and a symptomatic epiretinal membrane in the fellow eye; and one had bilateral POAG and congenital convergent strabismus.
- Healthy Volunteers: Fifteen healthy volunteers with no self-reported history of ocular disease.
Period: Overall Study
Arm/Group | Retinal Disease | Glaucoma | Strabismus | Ocular Comorbidities | Healthy Volunteers
Started | 14 | 13 | 14 | 4 | 15
Completed | 14 | 13 | 14 | 4 | 15
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retinal Disease | Glaucoma | Strabismus | Ocular Comorbidities | Healthy Volunteers | Total
Number analyzed (Participants) | 14 | 13 | 14 | 4 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 10 | 1 | 12 | 32
  >=65 years | 10 | 8 | 4 | 3 | 3 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (11.4) | 64.1 (14.7) | 50.8 (19.1) | 70.5 (8.0) | 53.1 (11.2) | 60.3 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 7 | 2 | 9 | 31
  Male | 8 | 6 | 7 | 2 | 6 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14 | 13 | 14 | 4 | 15 | 60
Visual acuity (better eye) [Mean (Standard Deviation); unit: logMAR] | 0.35 (0.24) | 0.10 (0.12) | -0.04 (0.08) | 0.24 (0.42) | 0.01 (0.14) | 0.18 (0.25)
Visual acuity (worse eye) [Mean (Standard Deviation); unit: logMAR] | 0.68 (0.34) | 0.20 (0.12) | 0.24 (0.27) | 0.63 (0.53) | 0.02 (0.15) | 0.33 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Total Examination Time
Description: Total time for each participant to complete the binocular optical coherence tomography (OCT) examination was calculated.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Retinal Disease | Glaucoma | Strabismus | Ocular Comorbidities | Healthy Volunteers
Number analyzed (Participants) | 14 | 13 | 14 | 4 | 15
seconds | 728.6 [654.7 to 826.4] | 676.7 [626.4 to 747.7] | 707.6 [636.9 to 847.9] | 620.6 [598.1 to 753.7] | 637.8 [572.4 to 821.7]

2. Secondary Outcome: Number of Participants With Subjective Ratings ≥ 4 on Post-Test Questionnaire
Description: Participants rated ease of use, duration, and appeal on a 5-point Likert scale in a post-test questionnaire.
Time Frame: 6 months
Population: Results based on a post-test questionnaire. Participants rated ease of use (from 1 to 5: 1 = very difficult, 5 = very easy), duration (from 1 to 5: 1 = very long, 5 = very short), and appeal (from 1 to 5: 1 = very unappealing, 5 = very appealing) on a 5-point Likert scale.
Measure: Count of Participants; unit: Participants
Arm/Group | Retinal Disease | Glaucoma | Strabismus | Ocular Comorbidities | Healthy Volunteers
Number analyzed (Participants) | 14 | 13 | 14 | 4 | 15
Participants
  Rated ≥ 4 ease of use | 9 | 11 | 12 | 2 | 13
  Rated ≥ 4 duration | 10 | 7 | 8 | 1 | 8
  Rated ≥ 4 appeal | 13 | 11 | 12 | 3 | 13

3. Secondary Outcome: Number of Participants That Presented Gradable Data, by Examination Type
Description: To identify potential user errors, particularly those with a likelihood of generating erroneous examination findings (e.g., failure to comply with device instructions or errors in voice recognition).
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Retinal Disease | Glaucoma | Strabismus | Ocular Comorbidities | Healthy Volunteers
Number analyzed (Participants) | 14 | 13 | 14 | 4 | 15
Participants
  Anterior segment imaging | 14 | 13 | 14 | 4 | 14
  Posterior segment imaging | 12 | 12 | 12 | 3 | 13
  Vitreous imaging | 12 | 12 | 12 | 3 | 13
  Motility | 10 | 9 | 12 | 2 | 14
  Visual acuity | 13 | 12 | 13 | 4 | 15
  Suprathreshold perimetry | 13 | 12 | 14 | 4 | 15
  Pupillometry | 11 | 10 | 13 | 4 | 13

ADVERSE EVENTS:
Arm/Group | Retinal Disease | Glaucoma | Strabismus | Ocular Comorbidities | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/14 | 0/4 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/14 | 0/4 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No